CLINICAL TRIAL: NCT05642884
Title: Feasibility of a Prehabilitation Intervention Among Older Adults With Myeloma Receiving Autologous Stem Cell Transplant
Brief Title: Prehabilitation Feasibility Among Older Adults Undergoing Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noha Mohamed Sharafeldin (Other)
Collaborators: O'Neal Comprehensive Cancer Center at UAB (Unknown)
Responsible Party: Sponsor-Investigator, Noha Mohamed Sharafeldin, Principal Investigator; Assistant Professor of Medicine, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAB 2281; O'Neal Invests (Other: UAB O'Neal Comprehensive Cancer Center)
Record Dates: First submitted 2022-11-10; First posted 2022-12-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Autologous Stem Cell Transplant
MeSH Terms: conditions — Multiple Myeloma | interventions — Nutrition Policy

STUDY DESIGN:
Intervention Model Description: We plan to enroll a total of 30 patients, randomized 1:1 using permuted block algorithm stratified by sex and age (e.g. 60-70, >70y), into intervention arm (home based prehabilitation) vs an attention control (dietary counseling) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teleprehab (Experimental): The participants selected for the teleprehab arm will undergo a supervised 8-week multi-modal exercise program in a telehealth format (using doxy.me, a free telehealth platform) delivered by licensed physical or occupational therapists who have undergone cancer specific rehabilitation training within Select Medical's ReVital® cancer rehabilitation program. Participants will attend teleprehab sessions 2 times per week for a total of 16 sessions.
  Interventions: Other: Multi-modal Exercise Regimen; Behavioral: Dietary Guidelines
- Attention Control (Other): The participants randomized to the attention control arm will not undergo an exercise regimen, but will be contacted by the study staff on the phone once a week..
  Interventions: Behavioral: Dietary Guidelines

INTERVENTIONS:
Other: Multi-modal Exercise Regimen — Participants will undergo a total of 16 sessions over 8 weeks. Each therapy session will comprise of patient education, including facilitated goal planning, promotion of physical activity and safe exercise guideline, followed by 30 minutes of preferred aerobic activity such as walking or biking.
  Arms: Teleprehab
Behavioral: Dietary Guidelines — Participants will be contacted once a week to review dietary recommendations per the 2022 American Cancer Society guidelines for cancer survivors.

SUMMARY:
This is a pilot feasibility trial among older adults (≥60y) scheduled to undergo Autologous Stem Cell transplantation at UAB. Participants will be randomized into either a prehabilitation program or an attention control group before their transplant. The primary outcomes will be feasibility and secondary outcomes include changes in physical function at the time of transplant and at 12 weeks follow up.

DETAILED DESCRIPTION:
This is a pilot randomized trial of older adults 60y and above planned to undergo Autologous Stem Cell Transplant for Multiple Myeloma. Eligible participants will be randomized (like flipping a coin) to one of two study conditions: 1) an 8 week long home-based prehabilitation exercise program delivered using a telehealth format or 2) an 8-week long nutrition counseling (attention control group). Assessments will occur at baseline, post-intervention (during transplant) and at 12-weeks post-transplant. Investigators will assess the feasibility and acceptability of our program as well as preliminary impact of the program on physical functioning during these time-periods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Myeloma
* Scheduled for ASCT at UAB within 10 weeks of study enrollment
* age at ASCT ≥60y

Exclusion Criteria:

* at high risk for impending pathologic fracture using Mirels score

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Participation rate | 1 year
  Participation rate will be measured as the number of participants agreeing to participate in the study divided by total participants approached for the study.
Completion rate | 1 year
  Completion rate will be measured as the number of participants completing the study intervention phase (8 weeks) divided by the total number of participants starting the intervention.
Adherence rate | 1 year
  Adherence rate will be computed Number of participants attending at least 80% of the planned intervention sessions divided by the total number of participants initiating the intervention.
Acceptability | 1 year
  Acceptability of intervention will be measured using a) 9-item Theoretical Framework of Acceptability Questionnaire which measures participants perspectives on the acceptability of the study intervention. Responses are measured in a likert type scale. and b) a semi-structured interview that will be focused on gathering overall acceptability of the intervention to the participants. Interview questions will be focused on understanding participants perspectives using 7 different proposed constructs of acceptability, i.e affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness and self efficacy.

SECONDARY OUTCOMES:
Change in Lower Extremity Physical Function | 1 year
  Investigators will measure lower extremity physical function using the Short Physical Performance Battery Scores (SPPB, score 0-12; higher score indicates better physical function) and compare the difference in SPPB scores before and after intervention
Change in Functional Exercise Capacity | 1 year
  Investigators will measure functional exercise capacity using 6-minute walking distance (6MWD) and compare the difference in 6MWD before and after intervention
Change in mobility | 1 year
  Investigators will measure mobility of study participants using the 9-item life space questionnaire (LSQ; score range 0-120, higher scores indicate better mobility) and compare the difference in LSQ before and after intervention
Change in functional status | 1 year
  Investigators will measure functional status using the Older Americans Resources and Services (OARS) Activities of Daily Living and Instrumental Activities of Daily Living (ADL/IADL) compare the difference in ADL/IADL scores before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Kirklin Clinic of UAB Hospital, Birmingham, Alabama, United States